CLINICAL TRIAL: NCT03476564
Title: Effects of Pentoxifylline and Vitamin E on Pregnancy Rate in Infertile Women Treated by ICSI: A Randomized Clinical Trial
Brief Title: Effects of Pentoxifylline and Vitamin E on Pregnancy Rate in Infertile Women Treated by ICSI:
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Collaborators: El Galaa Teaching Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Amr Fayez, doctor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BenhaU1
Record Dates: First submitted 2018-03-02; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Infertility, Female
Keywords: assisted reproductive techniques
MeSH Terms: conditions — Infertility, Female | interventions — Pentoxifylline

STUDY DESIGN:
Intervention Model Description: Endometrial thickness will be measured on the day of the HCG prescription in both groups by one of the two attending physicians. Chemical pregnancy will be detected by serum beta-hCG analysis 14 days after embryo transfer and transvaginal ultrasound scan will be scheduled 2 weeks later to confirm the diagnosis of clinical pregnancy. The intervention group will receive pentoxifylline (Trental S.R.) 400 mg/BD plus vit E (PHARCO) 400 mg/BD 2 cycles before starting ICSI cycle and the medication will be continued until the beta-hCG becomes positive or the cycle is cancelled. The comparison group will not receive the above drugs. The main outcome measure will be clinical pregnancy rate.
Who Masked: Participant
Masking Description: Computer generated random number table will be used for randomization. Group assignments will be placed in sealed opaque sequentially numbered envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): intervention group will receive pentoxifylline (Trental S.R.) 400 mg/BD plus vit E (PHARCO) 400 mg/BD 2 cycles before starting ICSI cycle and the medication will be continued until the beta-hCG becomes positive or the cycle is cancelled.
  Interventions: Drug: pentoxifylline; Drug: Vit E
- comparison group (No Intervention): . The comparison group will not receive the above drugs. The main outcome measure will be clinical pregnancy rate.

INTERVENTIONS:
Drug: pentoxifylline — will be given 2 cycles before starting ICSI cycle and the medication will be continued until the beta-hCG becomes positive or the cycle is cancelled
  Other Names: Trental S.R. 400 mg/BD
  Arms: intervention group
Drug: Vit E — will be given 2 cycles before starting ICSI cycle and the medication will be continued until the beta-hCG becomes positive or the cycle is cancelled
  Other Names: Vit E PHARCO 400 mg/BD
  Arms: intervention group

SUMMARY:
Our findings will provide preliminary clinical evidence to suggest the new experimental treatment approaches, toward female factor infertility treatment with pentoxyfylline.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted on 140 infertile patients. The study is approved by the Ethical Committee of Benha obstetrics and Gynecology Department and will be initiated after achieving written consents of the participants. The study will include infertile patients under 39 years of age without a previous history of ICSI cycle. Exclusion criteria will be hypothalamic amenorrhea, drug reactions or complications, endometriosis and fibroids. Patients will be randomly divided into two equal groups. Computer generated random number table will be used for randomization. Group assignments will be placed in sealed opaque sequentially numbered envelopes. For each participant a questionnaire will be filled by the researchers. The questionnaire contained questions about age, duration of infertility, the type and cause of infertility. Data will be collected from questionnaires, clinical, laboratory notes and ultrasound reports. Endometrial thickness will be measured on the day of the HCG prescription in both groups by one of the two attending physicians. Chemical pregnancy will be detected by serum beta-hCG analysis 14 days after embryo transfer and transvaginal ultrasound scan will be scheduled 2 weeks later to confirm the diagnosis of clinical pregnancy. The intervention group will receive pentoxifylline (Trental S.R.) 400 mg/BD plus vit E (PHARCO) 400 mg/BD 2 cycles before starting ICSI cycle and the medication will be continued until the beta-hCG becomes positive or the cycle is cancelled. The comparison group will not receive the above drugs. The main outcome measure will be clinical pregnancy rate.

Sample size calculation Sample size was calculated using PASS® version 11 program, setting the type-1 error (α) at 0.05 and the power (1-β) at 0.8. Results from a previous study (Ashraf alesyan, 2009) showed that the incidence of pregnancy rate among ttt group was 57.1% while for control group it was 39.2%, with an effect size of 12%. Calculation according to these values produced a minimal sample size of 131 cases in each group.

Results

Results will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* infertile female patients under 39 years

Exclusion Criteria:

* hypothalamic amenorrhea
* drug reactions or complications
* endometrioses
* fibroids

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female patients according to physical appearance and sex accepted socially
Enrollment: 140 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate. | two weeks after embryo transfer
  serum beta-hCG analysis 14 days after embryo transfer
clinical pregnancy rate | two weeks after embryo transfer
  transvaginal ultrasound scan will be scheduled 2 weeks after embryo transfer to confirm the diagnosis of clinical pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- El Galaa Teaching hosptial, Cairo, Ghamra, Egypt